CLINICAL TRIAL: NCT01609985
Title: Cutaneous Heart Sounds Data Collection During CRT Optimization Study
Brief Title: Cutaneous Heart Sounds Data Collection During Cardiac Resynchronization Therapy (CRT) Optimization Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Heart Sounds During CRT
Record Dates: First submitted 2012-03-28; First posted 2012-06-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy Defibrillator (CRT-D) Devices
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Cutaneous Heart Sounds Data Collection During CRT Optimization study is an acute, prospective, non-randomized multi-center feasibility clinical trial. The purpose of this clinical trial is to collect data to assist in the testing and finalization of a hemodynamic sensor-based cardiac resynchronization therapy (CRT) optimization scheme.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been implanted with a Medtronic market approved CRT-D device (Concerto®, Concerto® II, Maximo® II, Consulta®, Protecta™, or Protecta™ XT) within two years
* Subject must be 18 years of age or older
* Subject or his/her legally authorized representative has signed and dated the study specific informed consent form ("Consent Form")
* Subject is willing and able to comply with protocol requirements

Exclusion Criteria:

* Subject with atrial tachyarrhythmia or frequent atrial or ventricular ectopy
* Subject is post mitral or aortic valve repair or replacement
* Subject is participating in other research studies that many confound the results of this study
* Subject is pregnant or in fertile age without secure birth control
* Subject has dementia
* Subject is unwilling to comply with protocol requirements
* Subject has a device and lead system with fractured leads
* Subject cannot undergo an echocardiograph procedure, or is contraindicated to undergo such a procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with an implanted Medtronic market approved CRT-D device.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Collection of simultaneous cardiac signals representing heart sounds and CRT-D electrogram (EGM) vectors. | A two hour office visit within two years of CRT-Defibrillator (D) and lead system implant
  The cardiac signals collected by the modified Virtuoso® ICD and implanted CRT-D EGM vectors will be used to determine how to improve and finalize a prototyped hemodynamic sensor-based CRT optimization scheme.

SECONDARY OUTCOMES:
Comparison of modified Virtuoso® Implantable Cardiac Defibrillator (ICD) heart sounds and CRT-D electrogram (EGM) vectors | A two hour office visit within two years of CRT-D and lead system implant
  The heart sounds vector data from the externally affixed modified Virtuoso® ICD will be compared to the EGM vectors from the implanted CRT-D device after CRT optimization.
Determine if modified Virtuoso® ICD recorded heart sounds and CRT-D recorded EGM are able to detect phrenic nerve stimulation (PNS) | A two hour office visit within two years of CRT-D and lead system implant

CONTACTS AND LOCATIONS:
Overall Officials: Heart Sounds During CRT Clinical Trial Leader, Study Chair — Medtronic CRDM Clinical
Locations (5):
- United States (5):
  - Ronald Lo, Inc., Riverside, California
  - Orlando Health, Orlando, Florida
  - Essentia Institute of Rural Health, Duluth, Minnesota
  - Methodist DeBakey Cardiology Associates, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia